CLINICAL TRIAL: NCT02187809
Title: Multi-site, Prospective, Open-label, Long-term, Flexible Dose, Interventional Study to Evaluate the Safety and Tolerability of Clobazam as Adjunctive Therapy in Paediatric Patients Aged ≥1 to ≤16 Years With Dravet Syndrome
Brief Title: Safety and Tolerability of Clobazam as Adjunctive Therapy in Paediatric Patients Aged ≥1 to ≤16 Years With Dravet Syndrome
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to recruitment challenges
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14362B
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Results first posted 2017-02-15 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-02

CONDITIONS: Dravet Syndrome
MeSH Terms: conditions — Epilepsies, Myoclonic | interventions — Clobazam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clobazam (Experimental): A maximum of 2.0 mg/kg/day (maximum 80 mg/day) twice daily (BID); clobazam oral suspension (2.5 mg/mL) or clobazam scored tablets (10 mg), orally
  Interventions: Drug: Clobazam

INTERVENTIONS:
Drug: Clobazam
  Other Names: Onfi®

SUMMARY:
To investigate the long-term safety and tolerability of clobazam when administered for 1 year as adjunctive therapy in paediatric patients aged ≥1 to ≤16 years with Dravet Syndrome.

ELIGIBILITY:
The inclusion and exclusion criteria for the patients who participated in lead-in Study 14362A will be transferred from the 14362A study and for the patients who did not participate in lead-in Study 14362A the inclusion/exclusion is separately listed below.

Inclusion Criteria:

1. The patient has a diagnosis of Dravet Syndrome supported by:

   1. onset of seizures in the first year of life
   2. history of fever-induced prolonged seizures as determined by the Investigator

      * these may include prolonged (approximately 15 minutes or longer) hemi-clonic seizures
   3. multiple seizure types which may include:

      * generalised tonic-clonic (required for inclusion)
      * clonic (required for inclusion)
      * myoclonic jerks/seizures
   4. history of normal development prior to seizure onset followed by development delay or regression after seizure onset
   5. abnormal EEG consistent with Dravet Syndrome
2. The patient is currently receiving a stable dose of clobazam of at least 0.5 mg/kg/day (maximum 20 mg/day) for at least 3 months

Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (9):
- United States (8):
  - US010, Los Angeles, California
  - US012, Orange, California
  - US001, Orlando, Florida
  - US003, Rochester, Minnesota
  - US005, Kansas City, Missouri
  - US0011, Dallas, Texas
  - US006, Dallas, Texas
  - US004, Seattle, Washington
- MX003, Guadalajara, Mexico

RESULTS

PARTICIPANT FLOW:
Groups:
- Clobazam: A maximum of 2.0 mg/kg/day (maximum 80 mg/day) twice daily (BID); clobazam oral suspension (2.5 mg/mL) or clobazam scored tablets (10 mg), orally
  Clobazam
Period: Overall Study
Arm/Group | Clobazam
Started | 3
Treated | 1
Completed | 0
Not Completed | 3
Not completed — The study was terminated | 3

BASELINE CHARACTERISTICS:
Population: At the time of study termination, one patient had had been treated
Arm/Group | Clobazam
Number analyzed (Participants) | 1
Age, Continuous [Median (Full Range); unit: years] | 13 [13 to 13]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Time Frame: Up to Day 390
Population: At the time of study termination, only one patient had received IMP. No adverse events were observed in the study.
Measure: Number; unit: participants
Arm/Group | Clobazam
Number analyzed (Participants) | 1
participants | 0

2. Primary Outcome: Number of Participants With Adverse Events of Special Interest as a Measure of Safety and Tolerability Based on Dose
Time Frame: Up to Day 390
Population: At the time of study termination, only one patient had received IMP. No adverse events were observed in the study
Measure: Number; unit: participants
Arm/Group | Clobazam
Number analyzed (Participants) | 1
participants | 0

3. Primary Outcome: Columbia Suicide Severity Rating Scale (C-SSRS), Categorisation Based on Columbia Classification Algorithm of Suicide Assessment (C-CASA) Categories (1, 2, 3, 4 and 7) for Patients Aged ≥ 6 Years
Time Frame: Baseline and from Day 0 to Day 360
Population: At the time of study termination, one patient had received IMP. No C-SSRS data were collected from that single patient.
Arm/Group | Clobazam
Number analyzed (Participants) | 0

4. Primary Outcome: Change in Behavioural, Neurocognitive Measures Using Vineland Adaptive Behaviour Scale (VABS)
Time Frame: Baseline and from Day 0 to Day 360
Population: At the time of study termination, only one patient had received IMP. No VABS data were recorded for that single patient.
Arm/Group | Clobazam
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Mean Weekly Number of Tonic-clonic and Clonic Seizures
Time Frame: Baseline and from Day 0 to Day 360 and upon Study Completion/Withdrawal
Population: At the time of study termination, only one patient had received IMP. No seizure data were summarised for that single patient.
Arm/Group | Clobazam
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Initial Treatment Responders Who Returned to Their Baseline Tonic-clonic and Clonic Seizure Rate During the Study (an Assessment of Tachyphylaxis)
Time Frame: Baseline and from Day 0 to Day 360
Population: as for outcome 5
Arm/Group | Clobazam
Number analyzed (Participants) | 0

7. Secondary Outcome: Percentage of Initial Treatment Responders Who Returned to Their Baseline Tonic-clonic and Clonic Seizure Rate During the Study (an Assessment of Tachyphylaxis)
Time Frame: Baseline and from Day 0 to Day 360
Population: as for outcome 5
Arm/Group | Clobazam
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: One patient was treated for 33 days before study termination
Arm/Group | Clobazam
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects treated and no analysis. One patient was treated for 33 days.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No